CLINICAL TRIAL: NCT04140552
Title: Chinese Research Group of Gallbladder Cancer
Acronym: CRGGC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); Anhui Provincial Hospital (Other Government); The First Affiliated Hospital of Bengbu Medical University (Other); LanZhou University (Other); Henan Cancer Hospital (Other Government); The First Affiliated Hospital of Zhengzhou University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); Harbin Medical University (Other); The First Hospital of Jilin University (Other); Second Hospital of Jilin University (Other); China-Japan Union Hospital, Jilin University (Other); The First People's Hospital of Changzhou (Other); Changzhou No.2 People's Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China (Other); The First People's Hospital of Taicang (Unknown); Wuxi No. 2 People's Hospital (Other); Xuzhou Central Hospital (Other); Second Affiliated Hospital of Suzhou University (Other); Affiliated Hospital of Nantong University (Other); The First People's Hospital of Nantong (Unknown); The Affiliated Hospital of Xuzhou Medical University (Other); Second Affiliated Hospital of Nanchang University (Other); The First Affiliated Hospital of Nanchang University (Other); Jiangxi Provincial People's Hopital (Other); Shengjing Hospital (Other); Baotou Central Hospital (Other); Qinghai People's Hospital (Other); Changzhi Medical College (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Shanxi Provincial Cancer Hospital (Unknown); First Affiliated Hospital Xi'an Jiaotong University (Other); Eastern Hepatobiliary Surgery Hospital (Other); Shanghai Fengxian District Central Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Zhongshan Hospital (Other); Shanghai Pudong Hospital (Other); Central Hospital of Minhang District, Shanghai (Unknown); Putuo District People's Hospital of Shanghai (Unknown); Xinhua (Chongming) Hospital Affiliated to Shanghai Jiao Tong University School of Medicine (Unknown); Tianjin Medical University Cancer Hospital (Unknown); First Affiliated Hospital of Xinjiang Medical University (Other); First Affiliated Hospital of Kunming Medical University (Other); Yinzhou Hospital Affiliated to Medical School of Ningbo University (Other); Shaoxing Second Hospital (Other); Shaoxing People's Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Sir Run Run Shaw Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Zhejiang Cancer Hospital (Other); Huizhou Municipal Central Hospital (Other); Ningbo No. 1 Hospital (Other); People's Hospital of Hunan Province (Unknown); Hainan People's Hospital (Other); Taizhou Hospital (Other); Xinghua City People's Hospital (Unknown); Tongliao City Hospital (Unknown); Jiangxi Provincial Cancer Hospital (Other); Shandong Provincial Hospital (Other Government); Qilu Hospital of Shandong University (Other); The Affiliated Hospital of Qingdao University (Other); Xijing Hospital (Other)
Responsible Party: Principal Investigator, Yingbin Liu, MD, PhD, FACS, Prof., Shanghai Jiao Tong University School of Medicine
Other Study IDs: CRGGC_LYB_2019
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Gallbladder Neoplasms
Keywords: gallbladder neoplasms; gallbladder cancer
MeSH Terms: conditions — Gallbladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Chinese Research Group of Gallbladder Cancer (CRGGC) is a retrospective multicenter registry cohort, collecting electronic medical records of patients diagnosed with gallbladder cancer from hospitals in collaboration.

DETAILED DESCRIPTION:
The objectives of the CRGGC are as follows:

1. To study the current diagnosis and treatment of gallbladder cancer in China.
2. To clarify the prognostic role of debated risk factors associated with gallbladder cancer.
3. To improve the accurate staging of gallbladder cancer.
4. To standardize the treatment with gallbladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least clinical diagnosis of gallbladder cancer, including C23.9 and part of C24.0 (cystic duct cancer).
* Patients with accessible electronic medical record

Exclusion Criteria:

* Patients with undetermined primary site of cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from 2008 to 2020 diagnosed with gallbladder cancer in collaborated hospitals in China.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 5 years
  The overall survival data were defined by (date of death) - (date of first diagnosis). The survival status of patients were retrieved from follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Yingbin Liu, MD, PhD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (55):
- China (55):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Fifth Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - People's Hospital of Hunan Province, Changsha, Hunan
  - Baotou City Central Hospital, Baotou, Inner Mongolia
  - Changshu No.1 People's Hospital, Changshu, Jiangsu
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First People's Hospital of Nantong, Nantong, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The Second Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - The First People's Hospital of Taicang, Taicang, Jiangsu
  - Wuxi Second People's Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of Lanzhou University, Gansu, Lanzhou
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Qinghai Provincial People's Hospital, Xining, Qinghai
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Putuo District People's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital, Shanghai, Shanghai Municipality
  - Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality
  - Central Hospital of Minhang District, Shanghai, Shanghai Municipality
  - Shanghai Pudong Hospital, Shanghai, Shanghai Municipality
  - Shanghai Fengxian District Central Hospital, Shanghai, Shanghai Municipality
  - Xinhua (Chongming) Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The Second Affiliated Hospital of Zhejiang University School of medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Yinzhou Hospital Affiliated to Medical School of Ningbo University, Ningbo, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang
  - Shaoxing Second Hospital, Shaoxing, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
No plan for IPD access is scheduled.

REFERENCES:
- [Derived] Li L, Ren T, Liu K, Li ML, Geng YJ, Yang Y, Li HF, Li XC, Bao RF, Shu YJ, Weng H, Gong W, Lau WY, Wu XS, Liu YB. Development and Validation of a Prognostic Nomogram Based on the Systemic Immune-Inflammation Index for Resectable Gallbladder Cancer to Predict Survival and Chemotherapy Benefit. Front Oncol. 2021 Jun 29;11:692647. doi: 10.3389/fonc.2021.692647. eCollection 2021. PMID 34268122
- [Derived] Ren T, Li Y, Zhang X, Geng Y, Shao Z, Li M, Wu X, Wang XA, Liu F, Wu W, Shu Y, Bao R, Gong W, Dong P, Dang X, Liu C, Liu C, Sun B, Liu J, Wang L, Hong D, Qin R, Jiang X, Zhang X, Xu J, Jia J, Yang B, Li B, Dai C, Cao J, Cao H, Tao F, Zhang Z, Wang Y, Jin H, Cai H, Fei Z, Gu J, Han W, Feng X, Fang L, Zheng L, Zhu C, Wang K, Zhang X, Li X, Jin C, Qian Y, Cui Y, Xu Y, Wang X, Liu H, Hua Y, Liu C, Hao J, Wang C, Li Q, Li X, Liu J, Li M, Qiu Y, Wu B, Zheng J, Chen X, Zhu H, Hua K, Yan M, Wang P, Zang H, Ma X, Hong J, Liu Y. Protocol for a gallbladder cancer registry study in China: the Chinese Research Group of Gallbladder Cancer (CRGGC) study. BMJ Open. 2021 Feb 16;11(2):e038634. doi: 10.1136/bmjopen-2020-038634. PMID 33593763